CLINICAL TRIAL: NCT02788383
Title: Aplicación en la práctica clínica de la determinación Prenatal no Invasiva en el Genotipo RhD Fetal Durante el Primer Trimestre de la gestación en Gestantes RhD Negativas
Brief Title: Fetal RhD Genotye Non Invasive Prenatal Determination
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-RHD-2016-18
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Pregnant Women; Rh-Hr Blood-Group System

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Actually, our center is doing the prenatal determination of RhD fetal genotype in all RhD negative pregnant women.

The investigator want to demonstrate that this is an useful and efficient method.

DETAILED DESCRIPTION:
This is a retrospective observational study that pretend to demonstrate that the prenatal determination of RhD fetal genotype is useful and efficient in our clinical practice.

I'm going to check the clinical history of all negative RhD pregnant women since January 2013 until December 2015.

I'll check if prenatal determination matches with postnatal RhD determination of newborn.

Usually, when a RhD negative woman is pregnant we administrate gammaglobulin in 28 gestation weeks, after invasive procedures and after delivery if the baby is positive RhD.

Althought, the investigators know that the 40 percent of RhD negative pregnant have a negative RhD baby.

This study will do posible to know how many gammaglobulins hasn't been necessary thanks to prenatal determination.

This is an important thing because gammaglobulin is an humanoid product ( it isn't without heatlth risks,...) and because is expensive.

For this reason, if the investigators do universal determination of RhD fetal genotype the investigators can avoid the administration of humanoid product in pregnant women.

I want to demonstrate that this practice is very useful and efficient in our population.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant RhD negative women

Exclusion Criteria:

* Pregnant RhD positive women

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant RhD negative women since January 2013 until December 2015
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Prenatal determination fetal RhD genotype | Ten months
  RhD negative/ RhD positive

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided